CLINICAL TRIAL: NCT06680648
Title: Oxygen Insufflation Via a Flexible Scope to Remove Secretions and Blood Obstructiong the View When Advancing the Scope Towrds the Trachea
Brief Title: Oxygen Insufflation Via Flexible Scope
Acronym: OxyInsuffl
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Seltz Kristensen, Consultant anaesthesiologist, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OxygenInsufflation_F-24066560
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Insertion of a Flexible Bronchoscope; Airway Management When Secretions Obstruct the Larynx
Keywords: Flaxible Scope guided intubation; Fibreoptic intubation; The bleeding airway; The difficult airway

STUDY DESIGN:
Intervention Model Description: one arm is oxygen insufflation first followed by no-insufflation the second arm is: no insufflation followed by oxygen insufflation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insufflation first followed by no-insufflation (Experimental)
  Interventions: Procedure: addition of oxygeninsufflation via working channel of flexible scope
- no-insufflation first followed by insufflation (Active Comparator)
  Interventions: Procedure: no-oxygen insufflation

INTERVENTIONS:
Procedure: addition of oxygeninsufflation via working channel of flexible scope — addition of oxygeninsufflation via working channel of flexible scope in order to improve visibility when advancing the flexible scope
  Arms: Insufflation first followed by no-insufflation
Procedure: no-oxygen insufflation — no-oxygen insufflation added to the flexible scope while advancing it
  Arms: no-insufflation first followed by insufflation

SUMMARY:
The investigators will study to what extent insufflation of oxygen via the suction channel of a flexible bronchoscope can help with making access from the mouth to the trachea easier when there is blood or secretions in the way. We provide the oxygen-flow from the circle-system of an anaesthesia-machine and in this way we can limit the pressure to 30 and 40 cm H2O which are relatively safe pressure-levels. The endoscopy is performed on a plastic manikin and artificial sputum mixed with artificial blood is used. The procedure will be performed by 64 anaesthetists that will be randomised to use either oxygen-insufflation or not. The setup is cross-randomised so that each participant will perform two attempts, one with insufflation and one without. The procedures will be video-taped and evaluated by a blinded observer regarding a) success/failure of advancing the scope to the mid trachea under vision, b) the duration of the procedure. Additionally, subjective scores regarding the benefit of using insufflation will be obtained

DETAILED DESCRIPTION:
The investigators will study to what extent insufflation of oxygen via the suction channel of a flexible bronchoscope can help with making access from the mouth to the trachea easier when there is blood or secretions in the way. We provide the oxygen-flow from the circle-system of an anaesthesia-machine and in this way we can limit the pressure to 30 and 40 cm H2O which are relatively safe pressure-levels. The endoscopy is performed on a plastic manikin and artificial sputum mixed with artificial blood is used. The procedure will be performed by 64 anaesthetists that will be randomised to use either oxygen-insufflation or not. The setup is cross-randomised so that each participant will perform two attempts, one with insufflation and one without. The procedures will be video-taped and evaluated by a blinded observer regarding a) success/failure of advancing the scope to the mid trachea under vision, b) the duration of the procedure. Additionally, subjective scores regarding the benefit of using insufflation will be obtained

ELIGIBILITY:
Inclusion Criteria:

Anesthesiologists attending the airway course "Airwaymanagement for Anaesthesiologists"

-

Exclusion Criteria:

* non acceptance of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The fraction of bronchoscopic advancements that result in a view of vocal cords (Fully or partial) without the view being obstructed by saliva or blood during the advancement | 90 seconds
  The fraction in whom The flexible scope is advanced to the trachea with maintained visibility all the time until vocal cord is seen

SECONDARY OUTCOMES:
The scope is advanced to the trachea within 2 minutes | 2 minutes
  The flexible scope is advanced to the trachea with or without maintained visibility
Duration until the tip of the scope is in the trachea | 0-2 minutes
  Time from the tip of the scope passes the teeth until it is in the trachea
Operation percieved ease of advancing the scope to the trachea with maintained visibility | 2 minutes
  Operation percieved ease of advancing the scope to the trachea with maintained visibility, on a visual analogue scale from 1-10, 1 = very easy, 10 = almost impossible, lowest is best
Operation percieved ease of advancing the scope to the trachea, overall | 2 minute
  Operation percieved ease of advancing the scope to the trachea overall,
  , on a visual analogue scale from 1-10, 1 = very easy, 10 = almost impossible, lower score is best.
The scope is advanced to the trachea within 1 minute | 1 minute
  The flexible scope is advanced to the trachea with or without maintained visibility
unobstructed advancement to the trachea in two minutes | 2 minute
  The flexible scope is advanced to the trachea with maintained visibility
unobstructed advancement to the trachea in 90 seconds | 90 seconds
  The flexible scope is advanced to the trachea with maintained visibility
Obtaining a view of vocal cord(s) without obstruction of the view, obtained in 30 seconds | 30 sekunds
  The fraction of participants in each group who obtain a view of vocal cord(s) without the view being obstructed at any point
Obtaining a view of vocal cord(s) without obstruction of the view, obtained in one minute | 1 minute
  The fraction of participants in each group who obtain a view of the vocal cord(s) without the view being obstructed at any point
Obtaining a view of the vocal cord(s) without obstruction of the view, obtained in 90 seconds | 90 seconds
  The fraction of particip in each group who obtain a view of the vocal cord(s) without the view being obstructed, Obtained in 90 seconds
The fraction of brochoscopic advancements that results in Unobstructed advancement to the trachea in one minute | 1 minute
  The fraction of the attempts when the flexible scope is advanced to the trachea with maintained visibility

OTHER OUTCOMES:
Operator pecieved benefit of the addition of oxygen insufflation | 2 minutes
  After having tried the technique, the operator answers the question: How do you find that the addition of oxygen affects the advancement of the scope to the trachea? The aswer is on a VAS (Visual Analogue Scale) sale form -5 = "It makes it much worse" via "0" = neutral" to +5 ("it makes it much better"), higher is best

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Unoversity Hospital of Copenhagen, Copenhagen, The Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garioud A, Kristensen MS. Oxygen insufflation via the working channel during tracheal intubation guided by a flexible optical scope and benefits, dangers, and future of the method: a narrative review. BJA Open. 2024 Oct 17;12:100346. doi: 10.1016/j.bjao.2024.100346. eCollection 2024 Dec. PMID 39469423